CLINICAL TRIAL: NCT06096545
Title: Axillary Management After Neoadjuvant Chemotherapy: May Axillary Biopsy Replace Sentinel Lymph Node Biopsy?
Brief Title: Axillary Management After Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pelin Basım, Primary researcher, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Medipol Hospital 1
Record Dates: First submitted 2023-07-18; First posted 2023-10-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female
Keywords: locally advanced breast cancer; axillary involvement; neoadjuvant chemotherapy; axillary biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two groups based on the initial biopsy method. In Group A, patients with axillary metastasis identified by FNAB were subjected to repeat ultrasound-guided FNAB after completion of neoadjuvant treatment, while in Group B, patients with axillary metastasis identified by CNB underwent repeat biopsy using the same method after completing neoadjuvant treatment. The obtained biopsies were sent for histopathological evaluation without revealing patient names to avoid influencing the research results, and the surgical team was not informed of the biopsy results. During surgery, both dyed lymph nodes and clipped lymph nodes were excised for SLNB and assessed by frozen section evaluation. Thus, the predictability of axillary metastasis by preoperative FNAB/CNB was tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 = Fine needle aspiration biopsy (Active Comparator): In Group A, patients with axillary metastasis identified by FNAB were subjected to repeat ultrasound-guided FNAB after completion of neoadjuvant treatment, The obtained biopsies were sent for histopathological evaluation without revealing patient names to avoid influencing the research results, and the surgical team was not informed of the biopsy results. During surgery, both dyed lymph nodes and clipped lymph nodes were excised for SLNB and assessed by frozen section evaluation.
  Interventions: Procedure: Axillary sentinal lymph node biopsy
- Group 2 = Core biopsy (Active Comparator): in Group B, patients with axillary metastasis identified by CNB underwent repeat biopsy using the same method after completing neoadjuvant treatment.The obtained biopsies were sent for histopathological evaluation without revealing patient names to avoid influencing the research results, and the surgical team was not informed of the biopsy results. During surgery, both dyed lymph nodes and clipped lymph nodes were excised for SLNB and assessed by frozen section evaluation.
  Interventions: Procedure: Axillary sentinal lymph node biopsy

INTERVENTIONS:
Procedure: Axillary sentinal lymph node biopsy — For SLNB evaluation, multiple sections of the excised lymph node were stained with hematoxylin and eosin (H&E) at a thickness greater than 2 mm. Lymph nodes with metastasis greater than 2 mm were defined as positive SLNB. Macroscopic metastasis was considered positive in the evaluation for the axilla, while benign histological characteristics were considered negative. The presence of micrometastasis and isolated tumor cells was also noted. The size and diameter of the metastatic lymph node were considered in the evaluation.
  SLNB technique using isosulfan blue dye was performed for axillary evaluation, and all patients had the clipped lymph node excised under ultrasound guidance with a guide wire placed preoperatively.
  Other Names: Axillary dissection

SUMMARY:
The standard treatment for locally advanced and node-positive breast cancer is surgery following neoadjuvant chemotherapy (NAC). Using NAC in advanced-stage tumors and biologically aggressive subtypes can lead to de-escalation in surgical treatment for the breast and axilla.

Previously, NAC was believed to alter lymphatic drainage due to fibrosis and tumor emboli in lymphatic channels. However, the theAmerican College of Surgeons Oncology Group (ACOSOG) Z1071 and Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA) trials investigated the performance of sentinel lymph node biopsy (SLNB) after NAC in patients with proven axillary lymph node involvement at the initial biopsy.

In contemporary breast cancer management, particularly in the axillary approach, less invasive techniques are becoming increasingly common. This raises the question of whether there might be a patient group where SLNB could be avoided.

In this study, the investigators sought a new method to evaluate the axilla after NAC in patients with known axillary involvement previously. For this purpose, the investigators performed an ultrasound-guided needle biopsy on the clipped axillary lymph node with known metastasis before the planned surgery, aiming to assess the axilla without performing SLNB after treatment. Additionally, the investigators investigated which patient group might benefit more from this predictability based on molecular subtypes and clinical-pathological features.

DETAILED DESCRIPTION:
The current study was designed as a prospective randomized clinical trial conducted at two participating centers to evaluate the predictability of sentinel lymph node biopsy (SLNB) using axillary ultrasound-guided fine-needle aspiration biopsy (FNAB) and core needle biopsy (CNB) in patients with histologically proven axillary lymph node metastasis after neoadjuvant chemotherapy (NAC). The study was initiated after obtaining approval from the local ethics committee (Dated:06.03.3023/decision no:E-10840098-772.02-1685).

Patients:

Female patients aged 18 years and above with clinical stage T1-3 and biopsy-proven N1 breast cancer who received NAC were included in the study. Exclusion criteria were a history of axillary surgery or SLNB, prior axillary excisional lymph node surgery, N2-3 disease with a decision for initial axillary lymph node dissection (ALND), diagnosis of inflammatory breast cancer, presence of distant metastasis, incomplete chemotherapy, pregnancy, and lactation.

All participants underwent breast ultrasonography, mammography, and magnetic resonance imaging for imaging before NAC. Clipped lymph nodes that were histopathologically proven to be metastatic at the time of diagnosis underwent ultrasonography-guided CNB or FNAB seven days before surgery. Histopathological results after biopsy were grouped as negative, positive, and non-diagnostic for metastasis.

Patients were randomized into two groups based on the initial biopsy method. In Group A, patients with axillary metastasis identified by FNAB were subjected to repeat ultrasound-guided FNAB after completion of neoadjuvant treatment, while in Group B, patients with axillary metastasis identified by CNB underwent repeat biopsy using the same method after completing neoadjuvant treatment.

Surgical Technique and Nodal Evaluation:

SLNB technique using isosulfan blue dye was performed for axillary evaluation, and all patients had the clipped lymph node excised under ultrasound guidance with a guide wire placed preoperatively.

Inter-group Comparison:

Sensitivity, specificity, false-negative rate (FNR), false-positive rate (FPR), and accuracy values were compared between the two groups based on the needle biopsy and SLNB performed after NAC. In patients re-evaluated with FNAB and CNB after NAC, the effects of patient age, tumor size, radiological features of breast cancer and axillary lymph node, tumor and lymph node size, histopathological type and grade of tumor, receptor characteristics, maximum standardized uptake value (SUV) of the breast and axillary lymph node on Positron Emission Tomography and Computed Tomography (PET-CT), and differences in ER, PR, Her-2, and Ki 67 receptors in the final pathology were investigated on sensitivity, specificity, FNR, FPR, and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years-old female patients
* Clinical stage T1-3 and biopsy-proven N1 breast cancer
* Axillary nodal involvement
* Volunteer to participate in to study

Exclusion Criteria:

* A history of axillary surgery or SLNB, prior axillary excisional lymph node surgery,
* N2-3 disease with a decision for initial axillary lymph node dissection (ALND),
* Diagnosis of inflammatory breast cancer,
* Presence of distant metastasis
* Incomplete chemotherapy, pregnancy, and lactation
* T4 tumors
* Refusal to participate in to study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 50 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Prediction of axillary status after neoadjuvant chemotherapy without SLNB | through study completion, an average of 6 month
  In this study, the investigators sought a new method to evaluate the axilla after NAC in patients with known axillary involvement previously. For this purpose, the investigators performed an ultrasound-guided needle biopsy on the clipped axillary lymph node with known metastasis before the planned surgery, aiming to assess the axilla without performing SLNB after treatment.

SECONDARY OUTCOMES:
The investigators investigated which patient group might benefit more from this prediction based on molecular subtypes and the clinical-pathological features | through study completion, an average of 6 month
  Therefore, patient age, ultrasonographic parameters, maximum SUV of the breast and axillary lymph node on PET-CT, histopathological subtypes of breast cancer, largest tumor diameter, histopathological diagnosis, histological grade, estrogen, progesterone, Ki-67 and Her-2 receptor status will be evaluated and the effectiveness of these parameters in order to accurately assess the axillary lymph node without SLNB will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Basim, As. prof, MD, Principal Investigator — Medipol University / General Surgery Department; Emine YILDIRIM, As. prof, MD, Principal Investigator — Gaziosmanpasa Training and Research Hospital / General Surgery Department
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University Hospital, Istanbul, Bagcilar
  - Istanbul Gaziosmanpasa Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data

REFERENCES:
- [Background] You S, Kang DK, Jung YS, An YS, Jeon GS, Kim TH. Evaluation of lymph node status after neoadjuvant chemotherapy in breast cancer patients: comparison of diagnostic performance of ultrasound, MRI and (1)(8)F-FDG PET/CT. Br J Radiol. 2015 Aug;88(1052):20150143. doi: 10.1259/bjr.20150143. PMID 26110204
- [Background] Ha SM, Cha JH, Kim HH, Shin HJ, Chae EY, Choi WJ. Diagnostic performance of breast ultrasonography and MRI in the prediction of lymph node status after neoadjuvant chemotherapy for breast cancer. Acta Radiol. 2017 Oct;58(10):1198-1205. doi: 10.1177/0284185117690421. Epub 2017 Mar 28. PMID 28350255